CLINICAL TRIAL: NCT06877156
Title: Unipolar Signal Local Potential Measurement in Pulsed Field Ablation: A Pilot Study
Brief Title: Local Potential Measurement In PFA: A Pilot Study
Status: Completed | Type: Observational
Sponsor: CathVision ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: CVPFA-001
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- De Novo PFA ablation

SUMMARY:
This is a pilot study to collect unipolar signal data during a pulsed field ablation study for the treatment of atrial fibrillation and to test the performance of an algorithm designed to measure the local potential of the unipolar signal in real time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with paroxysmal or persistent atrial fibrillation (AF) undergoing first time PFA procedure indicated by investigator for the treatment of atrial fibrillation.

Male or non-pregnant female aged ≥18 years.

Able and willing to provide written informed consent prior to any clinical investigation related procedure

Exclusion Criteria:

* Pregnant or nursing subjects.
* Current participation in another investigational drug or device study that interferes with this study.
* Subjects who, in the opinion of the investigator, are not candidates for this study.
* Patients who have had a prior ablation procedure
* Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
* Life expectancy is less than 12 months, in the opinion of the investigator
* Subjects who, in the opinion of the investigator, are considered part of any vulnerable population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Paroxysmal and persistent atrial fibrillation patients referred for a cardiac ablation using pulsed field ablation.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2025-07-28 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
PFAnalyzer output | From enrollment to hospital discharge typically 1 day
  The automated peak-to-peak voltage of the local signal potential output from the PFAnalyzer will be compared to manual measurement of both unipolar and bipolar signals.

CONTACTS AND LOCATIONS:
Locations (1):
- KBC Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: Undecided